CLINICAL TRIAL: NCT06038786
Title: Resiliency Training on the College Campus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daphne Holt, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016P002351
Record Dates: First submitted 2023-08-28; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Psychotic Disorders; Mood Disorders; Anxiety Disorders
MeSH Terms: conditions — Psychotic Disorders; Mood Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Waitlist controlled design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resilience Training (Experimental): Participants obtained Resilience Training, a 4 session, 1.5 hour group intervention delivering the following skills: mindfulness, mentalization, and self-compassion.
  Interventions: Behavioral: Resilience Training
- Waitlist (Placebo Comparator): A 4-6 week waitlist during which participants did not receive any treatment. They would then obtain Resilience Training following their waitlist period.
  Interventions: Behavioral: Resilience Training

INTERVENTIONS:
Behavioral: Resilience Training — A 4 session group-based behavioral intervention which delivers the following skills: mindfulness, metallization, and self-compassion.

SUMMARY:
This is a waitlist controlled study examining the initial efficacy of Resilience Training among college students at an elevated risk for a severe mental illness.

ELIGIBILITY:
Inclusion Criteria:

1. 18-30 years old
2. Enrolled in undergraduate program at the college or university where the intervention takes place
3. Students who endorse delusion-like experiences (DLEs): Peter's et al. Delusion Inventory (PDI) score > 4 and/or
4. Students with mild to moderate depressive symptoms: Beck Depression Inventory (BDI) score ≥ 6

Exclusion Criteria:

1. Inability to provide informed consent
2. Not proficient in English
3. Current self-reported Diagnostic Statistical Manual 5 (DSM-5) diagnosis with active symptoms (such as active psychotic symptoms, current suicidality, serious active alcohol or substance use, marked deterioration in functioning over the prior month) determined by clinical interview with participant, or self-report of a psychiatric diagnosis that necessitates close monitoring or individual therapy and/or inpatient or partial hospitalization
4. Current enrollment in psychological or behavioral health treatment.
5. Current use of psychotropic medications (other than stimulants) prescribed by a physician.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Peters Delusions Inventory | Baseline, 4-weeks, 12 months
  The Peters Delusions Inventory (PDI) is a brief 21-item survey using non-stigmatizing and non-clinical language to obtain ratings of common delusional experiences (e.g. paranoia, grandiosity, ideas of reference) and perceptual aberrations (e.g. experiences of being controlled; thought insertion, withdrawal, and echoing). The PDI also captures conviction, preoccupation, and distress related to the delusions. This scale is scored from 0-21, with higher scores indicating more presence of these delusions.
Beck Depression Inventory | Baseline, 4-weeks, 12 months
  The Beck Depression Inventory (BDI) is a 21-item self-report assessment obtaining ratings of one's level of depression on a Likert scale of 0-63, with higher scores indicating more depressive symptoms.
Spielberger State-Trait Anxiety Inventory | Baseline, 4-weeks, 12 months
  The Spielberger State-Trait Anxiety Inventory (STAI) is a 20-item self-report scale obtaining ratings of one's anxiety, both those that are trait like and ongoing, and those that are state like and temporary. Scores range from 0-120, with higher scores indicate higher levels of anxiety symptoms.

SECONDARY OUTCOMES:
Connor-Davidson Resilience Scale | Baseline, 4-weeks, 12 months
  The Connor-Davidson Resilience Scale (CD-RISC) is a 25-item self-report scale obtaining ratings of one's level of coping and emotional resilience. It is rated on a scale of 0-100, with higher scores indicate one has more coping skills and more emotional resilience.
Five Facet Mindfulness Questionnaire | Baseline, 4-weeks, 12 months
  The Five Facet Mindfulness Questionnaire (FFMQ) is a 39-item self-report survey that obtains ratings of one's capacity for mindfulness. It contains 5 sub scales, although this study only used the total score. It is scored on a 0-195 scale, though a mean score is taken ranging from 0-5, with higher scores indicate greater capacity for mindfulness.
Interpersonal Reactivity Index | Baseline, 4-weeks, 12 months
  The Interpersonal Reactivity Index (IRI) is a 28-item self-report scale that measures one's ability to experience empathy for another person. The scale has 4 sub scales, yet this study utilized only two of them: the empathic concern and perspective taking subscales. It is scored on a 0-140 scale, with higher ratings indicate more ability for empathy.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Holt, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to submit the full, yet de-identified dataset to Mendeley Data: https://data.mendeley.com at publication of this manuscript.
Supporting Information: CSR, Analytic Code
Time Frame: Study data will be come available once manuscripts are published.
Access Criteria: Data shared will be coded, with no PHI included.
URL: http://data.mendeley.com

REFERENCES:
- [Derived] DeTore NR, Burke A, Nyer M, Holt DJ. A Brief Resilience-Enhancing Intervention and Loneliness in At-Risk Young Adults: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Feb 5;7(2):e2354728. doi: 10.1001/jamanetworkopen.2023.54728. PMID 38315488